CLINICAL TRIAL: NCT06640738
Title: Remifentanil and Dexmedetomidine in Uterine Fibroid Ablation: a Comparative Study
Brief Title: Investigating the Optimal Remifentanil and Dexmedetomidine Concentration for Uterine Fibroid Ablation
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Kaohsiung Medical University (Other)
Responsible Party: Principal Investigator, Tzu Ying Li, Attending Physician, Kaohsiung Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KMUHIRB-F(I)-20240227
Record Dates: First submitted 2024-09-27; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Uterine Fibroids (UF)
Keywords: Uterine Fibroids (UF); Remifentanil
MeSH Terms: conditions — Leiomyoma | interventions — DMAC2L protein, human

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- arm 1 (Experimental): During uterine fibroid ablation, the arm1 participant received Remifentanil [ ALVOGEN® (2 mg/vial)] 1.0 ng/mL via syringe infusion pump [Perfusor® Space | B. Braun] as a pain treatment.
  Interventions: Drug: arm 1
- arm 2 (Active Comparator): During uterine fibroid ablation, the arm2 participant received Remifentanil [ ALVOGEN® (2 mg/vial)] 2.0 ng/mL via syringe infusion pump [Perfusor® Space | B. Braun] as a pain treatment.
  Interventions: Drug: arm 2

INTERVENTIONS:
Drug: arm 2 — This study tries to find the best drug concentration of Remifentanil, ALVOGEN® (2 mg/vial) in Uterine Fibroid Ablation. We have two arms. Arm 1 with Remifentanil, ALVOGEN® (2 mg/vial) 1.0 ng/mL, and arm 2 with Remifentanil, ALVOGEN® (2 mg/vial) 2.0 ng/mL, both given via a syringe infusion pump, Perfusor® Space | B. Braun.
  Other Names: ALVOGEN; Remifentanil ALVOGEN®
  Arms: arm 2
Drug: arm 1 — This study tries to find the best drug concentration of Remifentanil, ALVOGEN® (2 mg/vial) in Uterine Fibroid Ablation. We have two arms. Arm 1 with Remifentanil, ALVOGEN® (2 mg/vial) 1.0 ng/mL, and arm 2 with Remifentanil, ALVOGEN® (2 mg/vial) 2.0 ng/mL, both given via a syringe infusion pump, Perfusor® Space | B. Braun.
  Other Names: Remifentanil ALVOGEN®
  Arms: arm 1

SUMMARY:
This clinical trial aims to find a better drug concentration of Remifentanil in Uterine Fibroid Ablation. The main question it seeks to answer is:

[primary hypothesis 1] Remifentanil concentration of 2.0 ng/mL provides better pain control in Uterine Fibroid Ablation.

There is a comparison group in this study: Researchers will compare Remifentanil concentration of 1.0 ng/mL to see if provides similar pain control with fewer side effects.

Participants will be separated into two groups, one group with a Remifentanil concentration of 2.0 ng/mL and the other 1.0 ng/mL. During uterine fibroid ablation, the patient's pain index will be recorded (using a Visual Analogue Scale (VAS) of 0~10 points). We will also record vital signs during the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 20 and 65 years old
* American Society of Anesthesiology classification I~III
* Female patients diagnosed with uterine fibroids by obstetricians and gynecologists

Exclusion Criteria:

1. Patients with heart disease (such as arrhythmia or severe ventricular dysfunction)
2. Patients with chronic kidney disease in stage III or above or dialysis patients
3. Long-term alcohol addiction or drug abuse
4. Patients with abnormal liver index or chronic hepatitis
5. Those who are allergic Remifentanil
6. Those who refuse to participate in the experiment

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Pain scores during uterine fibroid ablation | From the start of uterine fibroid ablation till 30 minutes after the ablation.
  Participants will be separated into 2 groups, one with remifentanil 1.0 ng/mL, and the other with remifentanil 2.0 ng/mL. Pain scores will be recorded during uterine fibroid ablation.

SECONDARY OUTCOMES:
Vital signs during uterine fibroid ablation | From the start of uterine fibroid ablation till 30 minutes after the ablation.
  Participants will be separated into 2 groups, one with remifentanil 1.0 ng/mL, and the other with remifentanil 2.0 ng/mL. Vital signs (including blood pressure, oxygen saturation and heart rates) will be recorded during uterine fibroid ablation.

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months and ending 3 years after the publication of results
Access Criteria: Researchers with a data sharing agreement may be able to share statistical Analysis Plan.